CLINICAL TRIAL: NCT07107113
Title: Pilates and Aerobic Training on Cardiorespiratory Fitness, Flexibility, Strength, and Muscular Power in Young Adults: a Randomized Controlled Clinical Trial
Brief Title: Pilates and Aerobic Training on Cardiorespiratory Fitness, Flexibility, Strength, and Muscular Power in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Raphael Goncalves de Oliveira, Professor, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GPASD_002_2025
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Improvement of Cardiorespiratory Fitness, Flexibility, Strength and Muscle Power in Healthy Participants
MeSH Terms: interventions — Exercise Movement Techniques; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilates (Experimental): A total of 13 exercises were selected for the Pilates group, including two stretching exercises and 11 strengthening exercises for the main muscle groups. Mat exercises and equipment exercises (Ladder Barrel, Cadillac, Step Chair, Reformer, Springboard, and Small Barrel) will be used. Two protocols will be adopted for progression (protocol 1: weeks 1-6; protocol 2: weeks 7-12). Two sets of 10 repetitions will be performed, with a 30-second rest between sets and exercises. The two-by-two rule will be used to increase the load. In this case, the load will increase when the participant performs ≥ 2 repetitions above their target of 10 repetitions in the last set, in two consecutive training sessions. The interventions will last 12 weeks, three times a week, for 60 minutes.
  Interventions: Other: Pilates Exercise
- Aerobic (Experimental): The aerobic group will perform walking/running exercises on a treadmill, using the extensive interval training method. To define the intensity and periodization of the training, the running speed associated with V̇O2max (vV̇O2max), second ventilatory threshold (vLV2), and average speed between vV̇O2max and vLV2 (v50%Δ) will be used as a reference. These parameters will be obtained from a maximal exercise test on a treadmill, performed before the start of the interventions. Two protocols will be adopted, with adjustments in density (work-to-recovery ratio) every two weeks. The interventions will last 12 weeks, three times a week, for 60 minutes.
  Interventions: Other: Aerobic exercises
- Pilates plus aerobic (Experimental): They will perform the same exercises as the Pilates group, however, with 1 set of 10 repetitions, with a 30-second rest between sets and exercises, totaling 30 minutes of intervention per session. In the second half of the intervention period, aerobic exercises will be performed, identical to those of the aerobic group, but for 30 minutes. The interventions will last 12 weeks, three times a week, for 60 minutes.
  Interventions: Other: Pilates exercises plus aerobic exercise
- Control (No Intervention): This group will be instructed to maintain their usual routine.

INTERVENTIONS:
Other: Pilates Exercise — Pilates exercises are characterized as muscle strengthening and stretching.
  Arms: Pilates
Other: Aerobic exercises — Aerobic exercises are characterized as a modality that works cardiorespiratory fitness.
  Arms: Aerobic
Other: Pilates exercises plus aerobic exercise — Pilates exercises are characterized as muscle strengthening and stretching, while aerobic exercises are characterized as a modality that works cardiorespiratory fitness.
  Arms: Pilates plus aerobic

SUMMARY:
Pilates exercises have been shown to be effective for a range of outcomes; however, it is unclear whether they can effectively contribute to improving cardiorespiratory fitness, especially when compared with aerobic training, which is known to be effective for this purpose. Furthermore, the differences between these modalities for outcomes such as flexibility, strength, and muscular power require further investigation. Therefore, the objective of this study is to assess the effectiveness of Pilates compared to aerobic training, as well as the combination of these activities, on cardiorespiratory fitness, flexibility, strength, and muscular power in young adults. Eighty women aged 18 to 40 will be randomized to four groups: Pilates (n = 20), aerobic (n = 20), Pilates plus aerobic (n = 20), and control (n = 20). Cardiorespiratory fitness will be assessed directly to estimate V̇O2max. Trunk flexibility in flexion and extension will be measured with a fleximeter (°). Lower-limb, upper-limb, and trunk muscle strength will be assessed by isokinetic dynamometry (N.m), while lower-limb muscle power (W) will be assessed by countermovement jumping on a force platform. Interventions will be conducted for 12 weeks, three times a week, with a 60-minute session duration. Analyses will be conducted by intention-to-treat and per-protocol.

ELIGIBILITY:
Inclusion Criteria:

* female;
* age between 18 and 40 years; - not having exercised in the last 6 months;
* agreeing not to perform any other type of exercise during the study period;
* being fit to exercise according to the Physical Activity Readiness Questionnaire (PAR-Q) criteria;
* having no musculoskeletal or neurological disorders that could affect exercise performance;
* having no known cardiovascular or respiratory diseases;
* having no cognitive impairment that could lead to the inability to follow simple commands;
* not being a smoker;
* not being pregnant;
* not being on any specific diets.

Exclusion Criteria:

* refusing to sign the informed consent form;
* being unable to complete the pre-intervention assessment procedures.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | Baseline and after 12 weeks
  Maximum volume of oxygen obtained directly from inhaled and exhaled gases (V̇O2max) in a maximum incremental treadmill test.

SECONDARY OUTCOMES:
Flexibility | Baseline and after 12 weeks
  Range of motion measured with a fleximeter (º) for trunk movement in flexion and extension.
Trunk muscle strength | Baseline and after 12 weeks
  Peak isokinetic torque of the trunk extensor and flexor muscles (cocentric/concentric) at 60°/s.
Lower limb muscle strength | Baseline and after 12 weeks
  Peak isokinetic torque of the knee extensor and flexor muscles (cocentric/concentric) at 60°/s.
Upper limb muscle strength | Baseline and after 12 weeks
  Peak isokinetic torque of the elbow extensor and flexor muscles (cocentric/concentric) at 60°/s.
Lower limb muscle power | Baseline and after 12 weeks
  Lower limb muscle power (W) measured by countermovement jump on a force plate.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be provided as supplementary material upon publication of the study results.
Supporting Information: SAP
Time Frame: From September 1, 2025, until the date of publication of the study.
Access Criteria: The information will be freely accessible.